CLINICAL TRIAL: NCT02329587
Title: tDCS for Inhibitory Control Deficits: A Test in OCD
Brief Title: Transcranial Direct Current Stimulation Augmented Exposure and Response Prevention for Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1405-003; 1R21MH104728-01 (NIH)
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERP plus tDCS (Experimental): ERP plus anodal tDCS of right inferior frontal gyrus
  Interventions: Other: ERP plus tDCS
- ERP plus sham tDCS (Active Comparator): ERP plus sham tDCS of right inferior frontal gyrus
  Interventions: Other: ERP plus sham tDCS

INTERVENTIONS:
Other: ERP plus tDCS — Participants in the ERP plus tDCS arm will receive an 11-session program, including 10 sessions which include both tDCS and ERP. During these sessions, 20 minutes of anodal tDCS will be delivered over right inferior frontal gyrus prior to the ERP exercise.
  Arms: ERP plus tDCS
Other: ERP plus sham tDCS — Participants in the ERP plus sham tDCS arm will receive an 11-session program, including 10 sessions which include both sham tDCS and ERP. During these sessions, 20 minutes of sham tDCS will be delivered over right inferior frontal gyrus prior to the ERP exercise.
  Arms: ERP plus sham tDCS

SUMMARY:
This study is investigating whether combining noninvasive brain stimulation with behavior therapy can help to improve outcomes for obsessive-compulsive disorder (OCD). Exposure and response prevention (ERP) -- a specific type of behavior therapy -- is a first line treatment for OCD. This study will test whether a form of noninvasive brain stimulation called transcranial direct current stimulation (tDCS), can help ERP work better.

ELIGIBILITY:
Inclusion Criteria:

* Current primary OCD diagnosis and current Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) total score of ≥16
* 18-65 years of age
* Ability to speak, read, write, and understand English sufficiently well to complete study procedures and provide informed consent
* Right-handed
* No use of psychiatric medications or stable psychiatric medication use for a minimum of 6 week prior to study entry. Psychiatric medications will be limited to the following: serotonin reuptake inhibitors (SRI; including clomipramine), combination antidepressants (including bupropion and serotonin-norepinephrine reuptake inhibitors), buspirone, benzodiazepines, and/or stimulants
* Naive to tDCS

Exclusion Criteria:

* Active substance use disorder
* Lifetime diagnosis of psychotic or bipolar mood disorder
* Previous minimally adequate trial of ERP (e.g., at least 16 sessions including both therapist and self-directed exposure and response prevention)
* Therapy outside the study protocol which has evidence for efficacy with OCD during the study intervention period
* Active suicidal or homicidal ideation
* Organic brain disease or injury
* Any health problems that would interfere with study participation, including contraindications to tDCS (e.g., skin condition, mental implant in skull)
* Women who are pregnant or breastfeeding. All women participants of child-bearing age are required to have a negative pregnancy test prior to treatment, and must use medically acceptable birth control during study participation. Medically acceptable birth control includes: established oral, injected, implanted, or vaginal ring hormonal contraception, an intrauterine device (IUD), two barrier contraception methods (condom or occlusive cap with spermicidal foam/gel/film/cream/suppository), or having a vasectomized partner
* Use of anticonvulsant medications (including depakote, gabapentin, tegretol, dilantin, lamictal) and/or glutamate-acting agents (including n-acetylcysteine, riluzole, amantadine, memantine).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-01; Primary Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Greenberg, MD, PhD, Principal Investigator — Butler Hospital; Sarah Garnaat, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A baseline assessment was completed between participant enrollment and randomization. Withdrawal during the baseline assessment could result in enrolled participants not being assigned to a treatment group.
Groups:
- ERP Plus tDCS: Exposure and response prevention (ERP) plus anodal transcranial direct current stimulation (tDCS) of right inferior frontal gyrus
  ERP plus tDCS: Participants in the ERP plus tDCS arm will receive an 11-session program, including 10 sessions which include both tDCS and ERP. During these sessions, 20 minutes of anodal tDCS will be delivered over right inferior frontal gyrus prior to the ERP exercise.
- ERP Plus Sham tDCS: Exposure and response prevention (ERP) plus sham transcranial direct current stimulation (tDCS) of right inferior frontal gyrus
  ERP plus sham tDCS: Participants in the ERP plus sham tDCS arm will receive an 11-session program, including 10 sessions which include both sham tDCS and ERP. During these sessions, 20 minutes of sham tDCS will be delivered over right inferior frontal gyrus prior to the ERP exercise.
Period: Baseline Thru Post-treatment Assessment
Arm/Group | ERP Plus tDCS | ERP Plus Sham tDCS
Started | 5 | 7
Completed All Intervention Sessions | 3 | 4
Completed | 4 | 6
Not Completed | 1 | 1
Period: 1-month Follow-up
Arm/Group | ERP Plus tDCS | ERP Plus Sham tDCS
Started | 4 | 6
Completed | 4 | 5
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ERP Plus tDCS | ERP Plus Sham tDCS | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.00 (17.42) | 39.86 (11.35) | 39.08 (13.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 7 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Yale-Brown Obsessive-Compulsive Scale (Y-BOCS): Total Score [Mean (Standard Deviation); unit: units on a scale] — The Y-BOCS is a well-known measure of obsessive-compulsive disorder (OCD) symptom severity. Total scores can range from 0-40, with higher scores corresponding to greater severity of symptoms.
  units on a scale | 24.80 (6.50) | 25.29 (4.27) | 25.08 (5.04)

OUTCOME MEASURES:

1. Primary Outcome: Yale-Brown Obsessive Compulsive Scale (Y-BOCS): Total Score
Description: The Y-BOCS is a well-known measure for assessing OCD symptom severity. Total scores can range from 0-40, with higher scores corresponding to greater severity of symptoms.
Time Frame: Post-treatment (approximately 6.5 weeks post-baseline)
Population: All participants with available data at the outcome timepoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ERP Plus tDCS | ERP Plus Sham tDCS
Number analyzed (Participants) | 4 | 6
units on a scale | 15.5 (8.50) | 16.33 (3.78)
Statistical Analysis 1: Comparison: ERP Plus tDCS vs ERP Plus Sham tDCS; Test type: Other; Between-group effect size (Hedge's g) = 0.138

2. Primary Outcome: Client Satisfaction Questionnaire-8: Total Score
Description: The Client Satisfaction Questionnaire-8 is measure of client satisfaction. Scores can range from 8-32, with higher scores corresponding to greater satisfaction.
Time Frame: Post-treatment (approximately 6.5 weeks post-baseline)
Population: All participants with available data on outcome measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ERP Plus tDCS | ERP Plus Sham tDCS
Number analyzed (Participants) | 4 | 5
units on a scale | 29.04 (2.76) | 29.60 (2.51)
Statistical Analysis 1: Comparison: ERP Plus tDCS vs ERP Plus Sham tDCS; Test type: Other; Between-group effect size (Hedge's g) = -0.214

3. Primary Outcome: Rates of Session Completion
Description: Average number of intervention sessions completed
Time Frame: Approximately 6.5 weeks post-baseline
Measure: Mean (Full Range); unit: Sessions
Arm/Group | ERP Plus tDCS | ERP Plus Sham tDCS
Number analyzed (Participants) | 5 | 7
Sessions | 8.40 [1 to 11] | 8.43 [1 to 11]
Statistical Analysis 1: Comparison: ERP Plus tDCS vs ERP Plus Sham tDCS; Test type: Other; Between-groups effect size (Hedge's g) = -0.007

4. Secondary Outcome: Yale-Brown Obsessive-Compulsive Scale: Total Score
Description: as for outcome 1
Time Frame: 1-month follow up (Approximately 11 weeks after baseline assessment)
Population: All available data for participants who completed the 1-month follow-up assesment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ERP Plus tDCS | ERP Plus Sham tDCS
Number analyzed (Participants) | 4 | 5
units on a scale | 17.25 (8.18) | 16.20 (5.89)
Statistical Analysis 1: Comparison: ERP Plus tDCS vs ERP Plus Sham tDCS; Test type: Other; Between-group effect size (Hedge's g) = -0.151

5. Secondary Outcome: Client Satisfaction Questionnaire-8: Total Score
Description: as for outcome 2
Time Frame: 1-month follow up (Approximately 11 weeks after baseline assessment)
Population: All available data for participants who completed the 1-month follow-up assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ERP Plus tDCS | ERP Plus Sham tDCS
Number analyzed (Participants) | 4 | 5
units on a scale | 30.75 (1.26) | 28.00 (5.05)
Statistical Analysis 1: Comparison: ERP Plus tDCS vs ERP Plus Sham tDCS; Test type: Other; Between-groups effect size (Hedge's g) = 0.704

6. Secondary Outcome: Rates of Retention in Intervention
Description: Number of randomized participants who remained in the intervention phase of the study and completed all intervention sessions.
Time Frame: Approximately 6.5 weeks post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ERP Plus tDCS | ERP Plus Sham tDCS
Number analyzed (Participants) | 5 | 7
Participants | 3 | 4
Statistical Analysis 1: Comparison: ERP Plus tDCS vs ERP Plus Sham tDCS; Test type: Other; Odds Ratio (OR) = 1.125

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline assessment through 1-month follow-up assessment (approximately 11 weeks post-baseline).
Arm/Group | ERP Plus tDCS | ERP Plus Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 4/5 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ERP Plus tDCS (N=5) | ERP Plus Sham tDCS (N=7)
Trouble sleeping (Nervous system disorders) | 1 | 0
Nightmares or other sleep disturbance (Nervous system disorders) | 4 | 2
Feeling drowsy or sleepy (Nervous system disorders) | 1 | 2
Feeling nervous or hyper (Nervous system disorders) | 1 | 1
Weakness or Fatigue (Nervous system disorders) | 1 | 2
Irritable (Nervous system disorders) | 2 | 3
Poor memory (Nervous system disorders) | 2 | 2
Trouble concentrating (Nervous system disorders) | 1 | 1
Feeling strange or unreal (Nervous system disorders) | 1 | 1
Numbness or tingling (Nervous system disorders) | 1 | 0
Dizziness or faintness (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 2 | 2
Blurred vision (Nervous system disorders) | 2 | 1
Ringing in ears or trouble hearing (Nervous system disorders) | 2 | 2
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dry mouth (Nervous system disorders) | 1 | 2
Muscle twitching or movements (Nervous system disorders) | 1 | 1
Trouble sitting still (Nervous system disorders) | 0 | 2
Tremor or shakiness (Nervous system disorders) | 2 | 2
Poor coordination or unsteadiness (Nervous system disorders) | 1 | 2
Heartbeat rapid or pounding (General disorders) | 1 | 1
Trouble catching breath or hyperventilation (General disorders) | 1 | 0
Nausea or vomiting (Gastrointestinal disorders) | 1 | 1
Stomach or abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 1
Loss of sexual interest (Nervous system disorders) | 1 | 0
Sweating excessively (Nervous system disorders) | 1 | 0
Fluid retention or swelling (General disorders) | 1 | 0
Appetite increased (Nervous system disorders) | 0 | 2
Weight gain (Metabolism and nutrition disorders) | 0 | 1
Skin rash or allergy (Immune system disorders) | 4 | 1
Diminished mental acuity/sharpness (Nervous system disorders) | 1 | 2
Difficulties finding words (Nervous system disorders) | 3 | 0
Apathy/emotional indifference (Nervous system disorders) | 0 | 1
Dizziness when you stand up (Vascular disorders) | 0 | 2
Bruising (Blood and lymphatic system disorders) | 1 | 1
Hot flashes (Endocrine disorders) | 1 | 0
Clenching of teeth at night (Nervous system disorders) | 0 | 2
Unable to sit still (Nervous system disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT02329587/Prot_SAP_000.pdf